CLINICAL TRIAL: NCT01260649
Title: N-methyl-D-aspartate Antagonist (Ketamine) Augmentation of Electroconvulsive Treatment for Severe Major Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding to cover staff salary (clinician and research coordinator)
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Instructor HMS, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010P001672
Record Dates: First submitted 2010-12-07; First posted 2010-12-15 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: Electroconvulsive treatment; ketamine; Major Depression; Treatment-resistant Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Sodium Chloride; Anesthetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketamine (Experimental): ketamine (0.5 mg/kg) followed by anesthetic agent titrated to sedation and succinylcholine titrated to muscle relaxation Right unilateral ECT at 5-6x seizure threshold three times a week
  Interventions: Drug: ketamine; Procedure: ECT; Drug: Muscle Relaxant; Drug: Anesthetic Agents
- placebo (Placebo Comparator): IV saline, followed by anesthestic agent titrated to sedation and succinylcholine titrated to muscle relaxation.
  Right unilateral ECT at 5-6x seizure threshold three times a week
  Interventions: Other: IV Saline; Procedure: ECT; Drug: Muscle Relaxant; Drug: Anesthetic Agents

INTERVENTIONS:
Drug: ketamine — eligible patients will be randomly assigned to a double-blind administration of ketamine (0.5 mg/kg) or IV Saline, followed by the routine anesthetic agent and muscle relaxant. ECT will be administered as per standard of care
  Arms: ketamine
Other: IV Saline — eligible patients will be randomly assigned to a double-blind administration of ketamine (0.5 mg/kg) or IV Saline, followed by the routine anesthetic agent and muscle relaxant. ECT will be administered as per standard of care
  Arms: placebo
Procedure: ECT — ECT will be administered as per standard of care
Drug: Muscle Relaxant — All participant will receive routine course of muscle relaxant with ECT as per standard of care
Drug: Anesthetic Agents — All participant will receive routine course of anesthetic agents with ECT as per standard of care

SUMMARY:
Electroconvulsive therapy (ECT), is considered the most effective treatment for severe treatment resistant major depressive disorder (MDD), but it requires about 3 weeks of treatments and can cause considerable acute deficits in memory. It would be a major advance in treatment if ECT could work faster with fewer treatments and result in decrease incidence of memory problems. Ketamine is an excellent candidate for augmentation of ECT because of its acute effects on depression, its short half-life, and its safety profile when given at low doses. Ketamine is given as an infusion and could easily be incorporated into the routine management of patients undergoing ECT, but has never been evaluated prospectively in this context.

The investigators propose to assess the efficacy, feasibility, tolerability and safety of N-methyl-D-aspartate antagonist augmentation of ECT using ketamine.

DETAILED DESCRIPTION:
Aim #1: To assess the efficacy of ketamine augmentation in reducing time to remission of a major depressive episode (MDE).

Aim #2: To assess the efficacy of ketamine augmentation on ECT-related cognitive side effects.

Aim #3: To assess the feasibility, safety, and tolerability of ketamine augmentation of ECT.

Exploratory aim #4: We propose to assess the patterns of functional connectivity before, during and after ECT using standard clinical EEG to better characterize the effect of ECT and to correlate clinical effects with changes in EEG measurements.

Thirty (30) participants will be recruited over 24 months. Participants will be males and females, ages 18-60, with severe MDD (baseline score HAM_D-28 >= 20) deemed appropriate for ECT treatment by their treating physician, agreeing to receive ECT treatment as part of their clinical care, and able to provide informed consent.

Exclusion criteria are any other DSM-IV primary diagnoses including major depressive disorder with psychotic features, bipolar disorder, schizoaffective disorder, schizophrenia, dementia, any history of psychosis, substance use disorder (abuse or dependence with active use within the last 6 months), and any lifetime history of ketamine abuse or dependence, organic mental disorders, seizure disorder or chronic antiepileptic medications, severe or unstable medical illness, pregnancy.

Study procedures: eligible patients will be randomized to a double-blind administration of ketamine (0.5 mg/kg) or saline before the first three ECT treatments. Right Unilateral ECT (RUL-ECT) will be administered at 6 times the seizure threshold, using the d'Elia placement of the electrodes. Electroconvulsive therapy will be given 3 times per week, as per standard of care at MGH. Depression severity will be assessed weekly with the HAM-D 28 (the main outcome measure), administered by a clinician blinded to randomization.

The neuropsychological assessment battery is designed to include instruments sensitive to the cognitive impairment associated with depression in general and ECT treatment in particular will be repeated at baseline, at the end of acute treatment series and at 3 months follow-up.

Also patients will undergo repeated EEG monitoring, at baseline after one week of treatment and at follow up with the aim of possibly identifying EEG features associated with response.

ELIGIBILITY:
Inclusion Criteria:

1. males and females between the ages of 18-65,
2. DSM-IV diagnosis of Major Depressive Disorder (MDD), without psychotic features
3. HAM-D-28 score of 20 or higher
4. requiring ECT treatment as part of their psychiatric care Comorbid anxiety disorders (OCD, Generalized anxiety, panic disorder) will be allowed as long as the clinician administering the SCID believes that they are not the primary diagnosis.

Exclusion Criteria:

1. MDD with a score of <20 on the HAM-D 28,
2. Other DSM-IV primary diagnoses including major depressive disorder with psychotic features, bipolar disorder, schizoaffective disorder, schizophrenia, dementia
3. any history of psychosis
4. substance use disorder (abuse or dependence with active use within the last 6 months), and any lifetime history of ketamine abuse or dependence;
5. organic mental disorders;
6. seizure disorder or chronic antiepileptic medications;
7. severe or unstable medical illness, including history of closed head injury resulting in loss of consciousness, medical contraindication to anesthesia or to ECT (i.e. recent myocardial infarction, increased intracranial pressure)
8. current treatment with memantine
9. pregnancy, or females of reproductive age who are not using an accepted method of contraception (birth control pill, IUD, combination of barrier methods).
10. known hypersensitivity to ketamine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2012-10-26 (Actual); Study Completion 2012-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine: ketamine (0.5 mg/kg) followed by anesthetic agent titrated to sedation and succinylcholine titrated to muscle relaxation Right unilateral ECT at 5-6x seizure threshold three times a week
  ketamine: eligible patients will be randomly assigned to a double-blind administration of ketamine (0.5 mg/kg), followed by the routine anesthetic agent and muscle relaxant. ECT will be administered as per standard of care
- Placebo: IV saline, followed by anesthestic agent titrated to sedation and succinylcholine titrated to muscle relaxation.
  Right unilateral ECT at 5-6x seizure threshold three times a week
  ketamine: eligible patients will be randomly assigned to a double-blind administration of ketamine (0.5 mg/kg), followed by the routine anesthetic agent and muscle relaxant. ECT will be administered as per standard of care
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 8 | 9
Completed | 6 | 8
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.43 (15.62) | 48.75 (12.22) | 48.57 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale - 28
Description: HAMD will be administered at every ECT treatment.The HAM D 28 is a 28 item scale with scores ranging from 0 to 83, with 0 being no depression and 83 being high levels of depression symptoms.
  The change in HAM S score was determined by the difference of the HAM D score at the last ECT administration and the baseline HAM D score. A negative change score reflects a decreased HAM D score between the first and last ECT administration and therefore a reduction in depressive symptoms.
Time Frame: baseline, one month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 6 | 8
units on a scale | -17.50 (6.53) | -14.00 (14.20)

2. Secondary Outcome: Number of Participants With Cognitive Side Effects
Description: will compare the incidence of participants with memory deficits between groups, as determined by incidents of clinician reported cognitive adverse events
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 6 | 8
Participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Ketamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/8
Other Adverse Events (participants affected / at risk) | 2/6 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=6) | Placebo (N=8)
Racing Thoughts (Psychiatric disorders) | 0 (0) | 1 (1)
Body pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=6) | Placebo (N=8)
Fluid in right ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sedation (Psychiatric disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Short term memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2)
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased Blood sugar (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Numbness in feet and body (Nervous system disorders) | 1 (1) | 0 (0)
Heart pounding/tightness in chest (Cardiac disorders) | 1 (1) | 0 (0)
Tingling in feet (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No